CLINICAL TRIAL: NCT02293473
Title: The Impact of Multimodal Monitoring During Major Surgery on the Morbidity, Mortality and Duration of Hospital Stay in UMC Ljubljana
Brief Title: Surgical Outcome and Multimodal Monitoring - SOMM
Acronym: SOMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, prof. Vesna Novak Jankovic, MD PhD, prof. Vesna Novak Jankovic, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: SOMM
Record Dates: First submitted 2014-06-10; First posted 2014-11-18 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Complications
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protocol Group (Experimental): Using multimodal monitoring to optimise the patients' haemodynamic status, namely, the use of LiDCO Rapid, BIS-Bispectral Index Monitor and INVOS-Cerebral Oxygenation Monitor monitors to assess and "fine tune" the patient, as described in the study protocol in detail.
  Interventions: Device: LiDCO Rapid; Device: BIS-Bispectral Index Monitor; Device: INVOS-Cerebral Oxygenation Monitor
- Control Group (Active Comparator): Using current standard of care
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: LiDCO Rapid — LiDCO Rapid haemodynamic monitor
  Arms: Protocol Group
Device: BIS-Bispectral Index Monitor — Depth of anaesthesia
  Arms: Protocol Group
Device: INVOS-Cerebral Oxygenation Monitor — regional brain tissue oxygenation
  Arms: Protocol Group
Other: Standard of care — Using standard of care
  Arms: Control Group

SUMMARY:
This study is designed to test if measuring the depth of anaesthesia, brain tissue oxygenation and haemodynamic parameters and specially designed interventions according to the measurements can improve the outcome of high risk surgical patients undergoing major abdominal surgery.

DETAILED DESCRIPTION:
All patients will be visited by a member of our team a day prior to surgery to seek an informed consent and to answer any questions. A set of laboratory results (see below) will be sought.

A test (Mini Mental test) will be performed to evaluate patients' cognitive functions. Our patients are fasted.

I. PROTOCOL GROUP

Pre-induction After the insertion of an intravenous catheter all patients will receive premedication (midazolam (Dormicum®) 1-2mg iv) and an arterial catheter will be inserted under local anaesthesia. Thoracic epidural catheter will be inserted in left lateral decubitus position (intervertebral space Th 7-8, or Th 9-10 for low intestinal surgery) and test with 3 ml of 2% lidocaine (Xylocaine®) will be performed.

LiDCO Rapid® (haemodynamics), unilateral INVOS® (brain tissue oxygenation) and unilateral BIS® (depth of anaesthesia) monitors will be applied. Should there be pre-existing carotid stenosis, INVOS® sensor will be applied on the ipsilateral side. In case of pre-existing cerebral pathology, the INVOS® sensor will be applied to the contralateral side. Baseline values of nominal stroke index (SI), cardiac index (CI), BIS value, mean arterial pressure (MAP) and regional tissue oxygen saturation (rSO2) will be recorded. Basal rSO2 will be recorded prior to preoxygenation.

1. Since the patients are fasted, 250ml of balanced crystalloid solution will be administered pre-induction. These will include antibiotics solvents and other pre-induction intravenous therapy.

Induction:

* Anaesthesia will be commenced using slow infusions of fentanyl (Fentanyl®) (3-5mcg/kg) or sufentanyl (Sufenta®) (0,3-0,5mcg/kg), followed by either propofol (Propofol®) (1-2mg/kg) or etomidate (Etomidate®) (0,2mg/kg), rocuronium (Esmeron®) (0,6mg/kg).
* Intubation, nasogastric tube, urine catheter, central venous line if needed.

Anaesthesia maintenance

* Sevoflurane (Sevorane®) in oxygen/air mixture, titration of volatile anaesthetic (see below)
* Bolus (slowly in 5 minutes) of 10-15 ml levobupivacaine (Chirocaine®) 0.25 % epidurally, with supplementation of sufentanyl (Sufenta®) 15 mcg.
* Epidural block will be considered efficient if no supplemental analgesia is needed during surgery (analgesia level Th1-L2). Should the block be inefficient, the patient will be excluded from further study. 1-2 hours after epidural bolus of local anaesthetic, infusion with PCEA (Patient Controlled Epidural Analgesia) analgesia mixture (0.125% levobupivacaine (Chirocaine®) 200 ml, morphine 4 mg, clonidine (Catapressan®) 0.075 mg) will be started. Hypotension due to sympathetic block will be treated with 250 ml of colloids and with an infusion of phenylephrine.
* Muscle relaxation monitoring and rocuronium (Esmeron®) (10-20 mg) supplementation, if needed. All patients will receive an antiemetic (granisetron (Kytril®) 1 mg) during the operation.
* Lungs will be ventilated with a tidal volume of ≥8ml/kg ideal body weight at approximately 10 times per minute.
* After induction of anaesthesia we will assess MAP changes and relative contributions to it of:

  * Excessive depth of anaesthesia (BIS outside 40-55 range)
  * Stroke volume and heart rate
  * Fluid status (see below) Appropriate measures will be taken.

Intraoperatively:

The aim of all the actions described below is to maintain CI, MAP and SI within 80% of baseline values.

1. Anaesthesia will be adjusted to maintain BIS 40-55

1. At the time of epidural bolus of local anaesthetic, an infusion of phenylephrine 0,01% 10-20ml/h will be started.
2. Maintenance fluids 2-3ml/kg/h of Hartmann's solution. Loss of blood will be substituted with colloids/red blood cells. In case of SVV (Stroke Volume Variation) >10% and SI and CI >10% below the starting value, a fluid challenge will be performed as follows: approximately 3ml/kg of colloid over maximum of 5 minutes. The response will be monitored. (In case of heart arrhythmias, SVV cannot be used. Any clinical indication of hypovolaemia will be tested using the above described fluid challenge and the response in SI.)

<!-- -->

1. If there is a fall in SVV and an increase in SI of >10% and the SVV% still >10%, a second fluid challenge will be performed.
2. If there is a reduction in SVV after fluid challenge, but increase in nSI <10% - no additional fluids will be given but vasoactive drugs (ephedrine, dobutamine or phenylephrine.
3. Any bradycardia (heart rate <60bpm) will be treated with administration of atropine 0,5 - 1,0 mg intravenously.

   2. A fall in rSO2 in the absence of a fall in nCI or blood loss - ventilation will be adjusted so that the PaCO2 will be kept in the high normal range (5-5,5kPa).

   Blood gas analysis will be performed at 1h intervals. 3. A fall in rSO2 with blood loss - haemoglobin level will be checked, if below agreed values (see 4) - blood will be administered.

   4. Hemoglobin will be kept above 80 g/L. A fall in haemoglobin will be coped with blood transfusion (see also 3). Should CI still be more than 10% below the baseline value, fluids or inotropes (e.g. dobutamine) will be administered (see 1b).

   5. Temperature will be held in the range between 36 and 37°C.

   Analgesia:

   • Epidurally, as described above

   End of operation:

   Muscle block reversal with sugammadex (Bridion®) 2-4 mg/kg.

   Post-operatively:

   Patients will be transferred to postoperative recovery and thereafter to Abdominal Surgery high dependency units (HDUs). Patients will thereafter be transferred to the ward. Additional data will be gathered in the HDU and at the ward for both, protocol and control group - see below.

   II. CONTROL GROUP

   Preinduction -as in protocol group

   Blinded monitoring LiDCO, INVOS and BIS monitors will be connected as in the protocol group, but the attending anaesthesiologist will be blinded to the measurements.

   Induction:

   -as in protocol group

   Fluids 2 ml/kg/h of balanced fluids + fluid loss replacement

   Anaesthesia maintenance

   • Sevoflurane (Sevorane®) (MAC-minimal alveolar concentration=1) in air/oxygen mixture (FiO2 0.40).

   • Bolus (5 min) of 10- 15 ml levobupivacaine (Chirocaine®) 0.25 % epidurally, with supplementation of sufentanyl (Sufenta®) 15 mcg. Epidural block will be considered efficient if no supplemental analgesia is needed during operation (analgesia level Th1-L2). Should the block be inefficient, the patient will be excluded from further study. 1-2 hours after epidural bolus of local anaesthetic, continuous infusion of PCEA mixture (0.125% levobupivacaine (Chirocaine®) 200 ml, morphine 4 mg, clonidine (Catapressan®) 0.075 mg) will be started.
   * Hypotension due to sympathetic block will be treated with 250 ml of colloids and with an infusion of phenylephrine.
   * Muscle relaxation monitoring and vecuronium (Norcuron®) (2-4mg) or rocuronium (Esmeron®) (10-20 mg) supplementation, if needed. All patients will receive an antiemetic (granisetron (Kytril®) 1 mg) during operation.

   End of operation:

   Muscle block reversal with sugammadex (Bridion®) (2-4 mg/kg).

   Post-operatively:

   Patients will be transferred to postoperative recovery and thereafter to Abdominal Surgery HDUs. Patients will then be transferred to the ward. Additional data will be gathered in the HDU and at the ward for both, protocol and control group - see below.

   III. DATA GATHERING

   We will record the following values:

   Intraoperatively:

   1. BIS value 2. INVOS Value 3. CI, SV, MAP, PPV, SVV, HRV from LiDCORapid 4. Duration of surgery 5. Blood loss and fluids given, transfusion 6. Temperature hourly 7. Haemoglobin, glucose, lactate, PaCO2 levels hourly

   Laboratory:

   A day prior to surgery, immediately after surgery and then each day for the duration of the stay:

   Haemogram, Na, K, Cl, Ca, Mg, Glucose, creatinine, uric acid, AST, ALT, gamma-GT, LDH, bilirubin, haemostasis, troponin, arterial blood gasses (as long as the patient has an arterial line), lactate, CRP, PCT

   Postoperatively:

   - Length of stay

   - Length of stay in HDU

   - Re-admissions to HDU

   - Admissions to ICU

   - Wound healing (yes/no)

   - Re-operations

   - 30 day mortality

   - Complications (sepsis, pneumonia, acute respiratory infection, pleural effusion, myocardial infarction, pulmonary embolism, stroke, intra-abdominal infection, urinary infection…)

   - Cognitive function test 1 week after surgery

   Daily also:
   * Body temperature
   * MAP
   * HR
   * SpO2
   * Diuresis (for as long as the patient has a urinary catheter)

   POWER ANALYSIS Using Wilcox test, for a 2 day difference in length of stay, with power 0,8 and significance level 0,05 16 patients in each group are needed, for showing 1 day difference in LOS, 63 patients in each group are needed. Calculations are based on a small pilot study.

ELIGIBILITY:
Inclusion Criteria:

* stomach surgery
* Pancreas surgery
* Large intestinal resections
* High risk surgical patients (ASA /American Society of Anesthesiologists/ 2-3 )

Exclusion Criteria:

* Pregnant women
* Laparoscopic surgery
* Palliative procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Reduced hospital stay | after release from hospital, an expected average of 10 days after surgery
  We are trying to prove that the protocol group will have a reduced hospital stay of 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Vesna Novak Jankovic, MD, PhD, Principal Investigator — UMC Ljubljana
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Background] Weiser TG, Regenbogen SE, Thompson KD, Haynes AB, Lipsitz SR, Berry WR, Gawande AA. An estimation of the global volume of surgery: a modelling strategy based on available data. Lancet. 2008 Jul 12;372(9633):139-144. doi: 10.1016/S0140-6736(08)60878-8. Epub 2008 Jun 24. PMID 18582931
- [Background] Findlay G, Goodwin A, Protopappa K, Smith N, Mason M. Knowing the risk: a review of the peri-operative care of surgical patients. London: National confidental enquiry into patient outcome and death (NCEPOD); 2011
- [Background] Story DA, Leslie K, Myles PS, Fink M, Poustie SJ, Forbes A, Yap S, Beavis V, Kerridge R; REASON Investigators, Australian and New Zealand College of Anaesthetists Trials Group. Complications and mortality in older surgical patients in Australia and New Zealand (the REASON study): a multicentre, prospective, observational study. Anaesthesia. 2010 Oct;65(10):1022-30. doi: 10.1111/j.1365-2044.2010.06478.x. PMID 20731639
- [Background] Quality and Performance in the NHS: NHS Performance Indicators London: NHS Executive; 2000
- [Background] Monk TG, Saini V, Weldon BC, Sigl JC. Anesthetic management and one-year mortality after noncardiac surgery. Anesth Analg. 2005 Jan;100(1):4-10. doi: 10.1213/01.ANE.0000147519.82841.5E. PMID 15616043
- [Background] Pearse RM, Moreno RP, Bauer P, Pelosi P, Metnitz P, Spies C, Vallet B, Vincent JL, Hoeft A, Rhodes A; European Surgical Outcomes Study (EuSOS) group for the Trials groups of the European Society of Intensive Care Medicine and the European Society of Anaesthesiology. Mortality after surgery in Europe: a 7 day cohort study. Lancet. 2012 Sep 22;380(9847):1059-65. doi: 10.1016/S0140-6736(12)61148-9. PMID 22998715
- [Background] Sessler DI, Sigl JC, Kelley SD, Chamoun NG, Manberg PJ, Saager L, Kurz A, Greenwald S. Hospital stay and mortality are increased in patients having a "triple low" of low blood pressure, low bispectral index, and low minimum alveolar concentration of volatile anesthesia. Anesthesiology. 2012 Jun;116(6):1195-203. doi: 10.1097/ALN.0b013e31825683dc. PMID 22546967
- [Background] Pearse R, Dawson D, Fawcett J, Rhodes A, Grounds RM, Bennett ED. Early goal-directed therapy after major surgery reduces complications and duration of hospital stay. A randomised, controlled trial [ISRCTN38797445]. Crit Care. 2005;9(6):R687-93. doi: 10.1186/cc3887. Epub 2005 Nov 8. PMID 16356219
- [Background] Shoemaker WC, Appel PL, Kram HB, Waxman K, Lee TS. Prospective trial of supranormal values of survivors as therapeutic goals in high-risk surgical patients. Chest. 1988 Dec;94(6):1176-86. doi: 10.1378/chest.94.6.1176. PMID 3191758
- [Background] Green D, Paklet L. Latest developments in peri-operative monitoring of the high-risk major surgery patient. Int J Surg. 2010;8(2):90-9. doi: 10.1016/j.ijsu.2009.12.004. Epub 2010 Jan 14. PMID 20079469
- [Background] Wilson J, Woods I, Fawcett J, Whall R, Dibb W, Morris C, McManus E. Reducing the risk of major elective surgery: randomised controlled trial of preoperative optimisation of oxygen delivery. BMJ. 1999 Apr 24;318(7191):1099-103. doi: 10.1136/bmj.318.7191.1099. PMID 10213716
- [Background] Sandham JD, Hull RD, Brant RF, Knox L, Pineo GF, Doig CJ, Laporta DP, Viner S, Passerini L, Devitt H, Kirby A, Jacka M; Canadian Critical Care Clinical Trials Group. A randomized, controlled trial of the use of pulmonary-artery catheters in high-risk surgical patients. N Engl J Med. 2003 Jan 2;348(1):5-14. doi: 10.1056/NEJMoa021108. PMID 12510037
- [Background] Walsh SR, Tang T, Bass S, Gaunt ME. Doppler-guided intra-operative fluid management during major abdominal surgery: systematic review and meta-analysis. Int J Clin Pract. 2008 Mar;62(3):466-70. doi: 10.1111/j.1742-1241.2007.01516.x. Epub 2007 Nov 21. PMID 18031528
- [Background] Abbas SM, Hill AG. Systematic review of the literature for the use of oesophageal Doppler monitor for fluid replacement in major abdominal surgery. Anaesthesia. 2008 Jan;63(1):44-51. doi: 10.1111/j.1365-2044.2007.05233.x. PMID 18086070
- [Background] Gurgel ST, do Nascimento P Jr. Maintaining tissue perfusion in high-risk surgical patients: a systematic review of randomized clinical trials. Anesth Analg. 2011 Jun;112(6):1384-91. doi: 10.1213/ANE.0b013e3182055384. Epub 2010 Dec 14. PMID 21156979
- [Derived] Jenko M, Jerin A, Spindler Vesel A. Biomarkers of neuroinflammation in abdominal cancer surgery with optimised anaesthesia. Acta Chim Slov. 2025 Jan 4;72(1):45-51. doi: 10.17344/acsi.2024.8901. PMID 40109058
- See also: Collaborator — http://www.vrvis.at/